CLINICAL TRIAL: NCT02038140
Title: Prospective Post Market Clinical Follow-Up (PMCF) Study of the Zimmer® Trabecular Metal™ Total Ankle
Brief Title: Zimmer Trabecular Metal Total Ankle PMCF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSU2011-07E
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Degenerative Arthritis; Rheumatoid Arthritis; Post Traumatic Arthritis
Keywords: Primary Ankle Replacement; Total Ankle Arthroplasty; Total Ankle Replacement; Trabecular Metal Total Ankle
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid | interventions — Arthroplasty, Replacement, Ankle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zimmer TM Total Ankle System (Other): Primary or revision total ankle arthroplasty subjects that receive the Zimmer Trabecular Metal Total Ankle System
  Interventions: Device: Zimmer Trabecular Metal Total Ankle System

INTERVENTIONS:
Device: Zimmer Trabecular Metal Total Ankle System — Primary or revision total ankle replacement
  Other Names: Primary Ankle Replacement; Total Ankle Arthroplasty; Total Ankle Replacement

SUMMARY:
The primary objective of this study is to obtain implant survivorship and clinical outcome data for commercially available Zimmer Trabecular Metal Total Ankle implants used in primary or revision total ankle arthroplasty. The assessment will include implant survivorship and clinical performance measured by pain and function, quality of life data, radiographic parameters and survivorship.

DETAILED DESCRIPTION:
The study design is a prospective, multicenter, study of the commercially available Zimmer Trabecular Metal Ankle semiconstrained implants. The study will require each site to obtain Institutional Review Board approval prior to study enrollment. All potential study subjects will be required to participate in the Informed Consent Process.

All study subjects will undergo preoperative clinical evaluations prior to their primary or revision total ankle arthroplasty. The post-operative clinical and radiographic evaluations will be conducted at 6 weeks, 6 month, 1 year, 2, 3, 5, 7, and 10 years. Follow-up surveys will occur at 4, 6, 8, and 9 years.

ELIGIBILITY:
Inclusion Criteria:

* The patient is > 18 years of age
* The patient is skeletally mature
* The patient qualifies for primary or revision total ankle replacement based on physical exam and medical history including the following: degenerative arthritis, rheumatoid arthritis, post-traumatic arthritis.
* The patient is willing and able to provide written informed consent
* Patient is willing and able to cooperate in the required post-operative therapy
* The patient is willing and able to complete scheduled follow-up evaluations questionnaires as described in the Informed Consent
* The patient has participated in the Informed Consent process and has signed the Institutional Review Board/European Commission approved Informed Consent

Exclusion Criteria:

* The patient is: a prisoner, mentally incompetent or unable to understand what participation in the study entails, a known alcohol or drug abuser, anticipated to be non-compliant.
* The patient has one of the following compromising the affected limb: ankle arthrodesis with malleolar exeresis, severe neurological or vascular disease, loss of musculature or neuromuscular compromise, severe instability, maltracking or misalignment of the tibia and talus uncorrectable by surgery.
* The patient has a local/systemic infection that may affect the prosthetic joint
* The patient has a previous history of infection in the affected joint
* The patient is known to be pregnant
* The patient has insufficient bone stock or bone quality to fix the components (i.e. osteoporosis, Charcot's disease)
* The patient has a known sensitivity or allergic reaction to one or more of the implanted materials
* The patient is unwilling or unable to give consent or to comply with the follow-up program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-03; Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Survivorship | 10 years
  Survival of the implants after 10 years which is based on removal of the prosthesis and will be determined using the Kaplan Meier Method.

SECONDARY OUTCOMES:
American Orthopaedic Foot and Ankle Society Score | First 2 years
  Performance os the Zimmer Trabecular Metal Ankle after 2 years which is assessed by the AOFAS score.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, MS, Study Director — Zimmer Biomet
Locations (11):
- United States (5):
  - University California Davis, Sacramento, California
  - Orthopaedic Associates of Grand Rapids REI, Grand Rapids, Michigan
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - The Rothman Institute, Philadelphia, Pennsylvania
- UBC Providence Health Care Research Institute, Vancouver, British Columbia, Canada
- Turku University Hospital Finland, Turku, Finland
- Klinikverbund St. Antonius und St. Josef GmbH, Wuppertal, Germany
- Humanitas San Pio X, Milan, Milano MI, Italy
- Switzerland (2):
  - Inselspital-Stiftung Universitatsspital Bern, Bern
  - Spital StS AG, Thun

IPD SHARING:
Plan to Share IPD: No